CLINICAL TRIAL: NCT03850028
Title: Molecular Imaging of Zirconium-89-labeled Atezolizumab as a Tool to Investigate Atezolizumab Biodistribution in High-risk Diffuse Large B-cell Lymphoma
Brief Title: Molecular Imaging Using Radiolabeled Atezolizumab to Assess Atezolizumab Biodistribution in Lymphoma Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed prematurely because the accrual was not achieved
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Stichting Hemato-Oncologie voor Volwassenen Nederland (Other); Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Marcel Nijland, hematologist and priniciple investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201700599; 2017-003511-20 (EudraCT Number); NL63047.042.18 (Other: CCMO)
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B-Cell Lymphoma, Not Otherwise Specified
Keywords: high risk DLBCL; molecular imaging; 89Zr-atezolizumab-PET; PDL1 imaging
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Other): All study participants will be allocated to this arm (single-arm study). Study participants will undergo a maximum of 3 89Zr-atezolizumab PET scans.
  Interventions: Other: 89Zr-atezolizumab PET scans

INTERVENTIONS:
Other: 89Zr-atezolizumab PET scans — The anti-PDL1 antibody atezolizumab, labeled with Zirconium-89 (89Zr) will be used as a molecular imaging tracer for PET scanning.
  These 89Zr-atezolizumab PET scans will be performed before and after induction therapy (R-CHOP) and at suspected relapse during or after consolidation treatment with atezolizumab (treatment trial HOVON 151).

SUMMARY:
Molecular imaging can be used for the noninvasive assessment of biodistribution of monoclonal antibodies. Atezolizumab has previously successfully been labeled with the radionucleotide Zirconium-89 (89Zr) and studied in solid malignancies (NCT02453984). The results of atezolizumab biodistribution can help to get a better understanding of the response mechanisms, the relation with minimal residual disease, the relation with the status of the T-cell and natural killer (NK)-cell repertoire and toxicity of programmed death ligand 1 (PDL1) checkpoint inhibition. Possibly in the future this will facilitate optimal patient selection. Sequential 89Zr-atezolizumab positron emission tomography (PET) scans can provide information on the dynamics of atezolizumab biodistribution over time. In combination with repeated characterization of tumor tissue and blood samples, these results can give inside in primary and acquired resistance.

In this parallel study of the HOVON 151 trial, 89Zr-atezolizumab-PET-scans will be used to evaluate 20 high risk DLBCL patients before and after induction (R-CHOP) therapy, and at suspected relapse during or after atezolizumab consolidation (HOVON 151).

DETAILED DESCRIPTION:
Patients with a high risk diffuse large B-cell lymphoma (DLBLC) with an international prognostic score (IPI) > 2, have a high risk of relapse even after achieving a metabolic complete remission with cyclophosphamide, doxorubicin, vincristine, prednisone and rituximab (R-CHOP) chemo-immunotherapy. Outcome after relapse is dismal. In patients with varies types of relapsed lymphoma checkpoint inhibition have shown promising results.

In order to improve outcome patients with a high risk DLBCL will be treated in the HOVON 151 trial (EudracT 2017-002605-35) with the monoclonal antibody directed against the immune checkpoint program death ligand 1 (PDL1) atezolizumab for 1 year after achieving a complete metabolic remission with R-CHOP.

The observed percentage of PDL1 positive tumor cells in DLBCL cases ranges from 13 to 31%. For PD-1/PDL1 checkpoint inhibition PDL1 tumor surface expression was proposed as a potential predictive marker. Despite higher overall response rates in PDL1 positive malignancies compared to PDL1 negative tumors, responses are seen in PDL1 negative patients nevertheless. PDL1 status from resected specimens showed a poor correlation to the PDL1 status from matched biopsies. Furthermore it has been shown that PDL1 expression in tumor biopsies changes with treatment. Therefore, PDL1 expression assessed by one single biopsy might not be representative.

Molecular imaging can be used for the noninvasive assessment of biodistribution of monoclonal antibodies. Atezolizumab has previously successfully been labeled with the radionucleotide Zirconium-89 (89Zr) and studied in solid malignancies (NCT02453984). The results of atezolizumab biodistribution can help to get a better understanding of the response mechanisms, the relation with minimal residual disease, the relation with the status of the T-cell and natural killer (NK)-cell repertoire and toxicity of programmed death ligand 1 (PDL1) checkpoint inhibition. Possibly in the future this will facilitate optimal patient selections. Sequential 89Zr-atezolizumab PET scans can provide information on the dynamics of atezolizumab biodistribution over time. In combination with repeated characterization of tumor tissue and blood samples, these results can give inside in the primary and acquired resistance.

In this parallel study of the HOVON 151 trial, 89Zr-atezolizumab-PET-scans will be used to evaluate 20 high risk DLBCL patients before and after induction (R-CHOP) therapy, and at suspected relapse during or after atezolizumab consolidation (HOVON 151).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 (inclusive) years
* Patients with a confirmed histologic diagnosis of diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS) based upon a representative histology specimen according to the World Health Organization (WHO) classification, revision 2016 (see appendix A)
* Ann Arbor stages II-IV (see appendix B)
* WHO performance status 0 - 1 (see appendix E)
* international prognostic index (IPI) ≥ 3 at diagnosis (see appendix C)
* Negative pregnancy test at study entry
* Patient is willing and able use adequate contraception during and until 5 months after the last protocol treatment.
* Written informed consent
* Patient is capable of giving a written informed consent

Exclusion Criteria:

Diagnosis

* All histopathological diagnoses other than DLBCL-NOS according to the WHO classification, revision 2016 (see appendix A), including:
* High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 translocations
* Testicular large B-cell lymphoma
* Primary mediastinal B cell lymphoma
* Transformed indolent lymphoma
* Post-transplant lymphoproliferative disorder

Organ dysfunction

* Clinical signs of severe pulmonary dysfunction
* Clinical signs of heart failure (NYHA classification II-IV)
* Symptomatic coronary artery disease or cardiac arrhythmias not well controlled with medication.
* Myocardial infarction during the last 6 months
* Significant renal dysfunction (serum creatinine ≥ 150 umol/l or clearance ≤ 30ml/min

Creatinine clearance (CrCl) may be calculated by Cockcroft -Gault formula:

CrCl = (140 - age [in years]) x weight [kg] (x 0.85 for females) / (0.815 x serum creatinine [μmol/L])

* Inadequate hematological function: hemoglobin < 5.5 mmol/L,absolute neutrophil count (ANC) < 1.0x10^9/L or platelets < 75x10^9 /L
* Spontaneous international normalized ratio (INR) > 1.5, activated partial thromboplastin time (aPTT) >33
* Significant hepatic dysfunction (total bilirubin ≥ 1.5x upper limit of normal (ULN) or transaminases ≥ 2.5 x ULN), unless related to Gilberts syndrome.
* Clinical signs of severe cerebral dysfunction
* Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
* Major surgery within the last 4 weeks

Known or suspected infection

* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks before date of registration. Suspected active or latent tuberculosis needs to be confirmed by positive interferon gamma (IFN-γ) release assay
* Patients known to be human immunodeficiency virus (HIV)-positive
* Active chronic hepatitis B or C infection
* Administration of a live, attenuated vaccine within 4 weeks before date of registration or anticipation that such a live attenuated vaccine will be required during the study and for a period of 5 months after discontinuation of atezolizumab

Auto-immune

* Any active or history of documented autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. The following exceptions are allowed: Patients with autoimmune-related hypothyroidism or type 1 diabetes mellitus who are on stable treatment.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest CT scan at screening.
* Patients with uncontrolled asthma or allergy, requiring systemic steroid treatment
* Regular treatment with corticosteroids within the 4 weeks prior to date of registration, unless administered for indications other than non-Hodgkin lymphoma (NHL) at a dose equivalent to < 30 mg/day prednisone/prednisolone.

General

* Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease)
* Current participation in another clinical trial interfering with this trial
* History of active cancer during the past 5 years, except basal cell carcinoma of the skin or stage 0 cervical carcinoma
* Life expectancy < 6 months
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Prior treatment

* Prior treatment with atezolizumab, or anti PD1 or PDL1 antibodies.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) therapeutic antibodies.
* Treatment with systemic immunostimulatory agents (including but not limited to interferon (IFN), interleukin (IL)-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to date of registration.
* Treatment with systemic immunosuppressive medications, including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti- tumor necrosis factor (anti-TNF) agents within 2 weeks prior to date of registration; inhaled corticosteroids and mineralocorticoids are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 89Zr-atezolizumab | From 2 weeks before R-CHOP until 52 weeks after R-CHOP
  The biodistribution of the tracer 89Zr-atezolizumab as assessed with 89Zr-atezolizumab PET scans.

SECONDARY OUTCOMES:
PDL1 and human leukocyte antigen (HLA) expression using immunohistochemistry (IHC) | IHC for PDL1 and HLA expression on archival tumor tissue will be performed after initial biopsy at time of diagnosis.
  Tumor and immune cell PDL1 and HLA expression on archival pre-treatment biopsy via IHC.
Soluble programmed death ligand 1 (sPDL1) measurement using an enzyme-linked immunosorbent assay (ELISA). | From 2 weeks before R-CHOP until 52 weeks after R-CHOP
  sPDL1 serum levels will be determined with ELISA
Gene expression profiling (GEP) via Nanostring | From 2 weeks before R-CHOP until 52 weeks after R-CHOP
  GEP via Nanostring analysis for cell-of origin will be perfomed on archival, paraffin fixed biopsies.
Next generation sequencing (NGS) data | From 2 weeks before R-CHOP until 52 weeks after R-CHOP
  Mutational analysis will be perfomed on archival, paraffin fixed biopsies.

OTHER OUTCOMES:
T- and NK-cell dynamics in response to R-CHOP therapy | From 2 weeks before R-CHOP until 52 weeks after R-CHOP
  Multi-parameter flowcytometry will be used to assess baseline and post induction-therapy status of the T- and NK-cell repertoire.
Gut microbiome dynamics in response to R-CHOP therapy | From 2 weeks before R-CHOP until 52 weeks after R-CHOP
  Baseline and post induction-therapy fecal samples will be collected for NGS analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Nijland, MD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - VU University Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No